CLINICAL TRIAL: NCT02832414
Title: Effectiveness of an Intensive Weight Loss Program for Obstructive Sleep Apnea Syndrome (OSAS) Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Linde AG (Industry)
Responsible Party: Principal Investigator, Carmen Monasterio, Doctor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR209/14
Record Dates: First submitted 2016-07-06; First posted 2016-07-14 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea, Obstructive; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

ARMS (2):
- Regular program (No Intervention)
- Intensive weight loss program (Active Comparator)
  Interventions: Behavioral: Intensive weight loss program

INTERVENTIONS:
Behavioral: Intensive weight loss program — behavioral and dietary supplement
  Arms: Intensive weight loss program

SUMMARY:
The purpose of this study is to determine if a lifestyle change program for obese patients who are already receiving continuous positive airway pressure (CPAP) treatment can achieve weight loss and overall improvement of obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
Calculating the sample size:

The primary endpoint is the reduction of final apnea-hypopnea index (AHI) with respect to baseline. Assuming an alpha level of 0.05 and a bilateral approach to have 80% statistical power, the investigators estimate a final sample size of 42 patients is required to detect a 15 point difference in AHI between the intervention and control groups (clinically relevant difference), with a standard deviation of 15 (visit 9) and accounting for a 25% rate of attrition. Balanced groups are expected.

Lifestyle Change Program:

This will consist of a 3-month long first stage of intensive diet and progressive exercise with visits to a nutritionist every 15 days. A second stage will last until completion of one year, with a diet that is progressively higher in calories, more intense exercise, appointments that are spaced further apart and are alternatively individual and group visits.

Diet First stage: 12 weeks

1. first 15 days: Very low calorie diet. A diet that is very low in calories will be started (600-800 kilocalories (Kcal), based on gender and level of physical activity) with low calorie shakes. Supplementing the diet with herbal teas and sugar-free beverages will be allowed.
2. Up to week 12: 1200 Kcal diet with a low calorie shake replacing the evening meal. Exercising begins.

At each visit the nutritionist will provide advice on diet and lifestyle, with special emphasis on diet and exercise. Visits to the nutritionist will be every 15 days. The first two will be group visits and afterwards individual visits will alternate with group visits every 15 days (see chart below). On alternate weeks a nurse will phone the patients to remind them of the diet's basic guidelines.

Every session will last from 60 to 90 minutes and will be conducted by a nutritionist. The subjects will be asked to keep a 3 day log of what they eat at the start of the study and at and at each visit in order to estimate nutrient intake. Every patient will be provided with information about the entire program and the different group and individual sessions with the nutritionist. At each visit the participants will be weighed and asked for the results of the tests for ketones in the urine once a week. The nutritionist will follow compliance with the program and monitor for potential adverse events at each visit.

Second stage: from 12 weeks to 1 year A 1200-1500 Kcal diet will be maintained, based on gender and level of physical activity, without the low calorie shake. Calorie intake will be based on a Mediterranean diet, recommending a maximum fat intake of 30% and high consumption of fruit, vegetables, poultry, fish, lean meat and legumes, in accordance with the recommendations of the American Dietetic Association.

Visits to the nutritionist will take place monthly from the third to the sixth month and every 3 months from the sixth to the 12th month, with individual visits alternating with group visits (see chart below).

They will also receive a phone call every month, alternating with the visits, which will be made by the company that supplies the CPAP equipment.

Exercise

The following exercise program will be recommended:

1. Walk briskly for at least 50-60 minutes at a time, at least 3 times per week, ideally 5 days a week. Exercising is to increase gradually, starting with 10 minute periods, repeated on the same day and that will be gradually increased as tolerated by the patient. Heart rate will be used to monitor exercise intensity, it is recommended that aerobic exercise be performed at 70-80% of maximum heart rate. (Lung (2014) 192:175-184).
2. Every workout session will consist of stretching, 5-10' of warm up (50-60% of maximum heart rate (HR)), 40-50' of aerobic exercise performed at 70-80% of maximum HR and 5-10' of cool down (50-60% of maximum HR). The table for stretches to be performed before and after exercising will be given in writing. The patients will receive information on how to perform the exercises and everything related to it at a group training session before the start of the program.
3. To encourage exercise, the chance to perform it at least once a week in guided groups, in the patient's town of residence, will be offered.

Follow up:

1. On each visit to the nutritionist, in addition to data regarding adherence to the diet, data regarding adherence to the exercise program will be recorded: number of sessions and minutes/week.
2. During the group sessions, the nurse in charge of the study will respond any questions that may arise concerning the development of the exercise program.
3. Patients who have a smart phone will also be able to record their activity using an app (Endomondo) , which the nurse and the nutritionist will be able to access (see the section on variables). In addition to tracking their own exercise history, patients will be able to see that of the other patients in the study if they opt voluntarily to choose that option.

If any musculoskeletal complaints that are deemed relevant should occur during the course of the exercise program, the Rehabilitation Services will attend to the patients. The pain visual analogue scale (VAS) will be used for assessment. A VAS score equal to or greater than 4 (moderate pain) would require assessment to be made by the Rehabilitation Services.

Assessment of exercise capacity:

1 To measure the response to exercise an exercise tolerance test will be performed: the six minute walk test (6MWT), which will be evaluated using the reference values for obese individuals. It will be conducted before starting the program and at 3 and 12 months.

Sleep habits Subjects will be reminded of the need to sleep enough hours and of keeping a regular sleep schedule. Sleep hygiene guidelines will be provided in writing.

Control group: They will be managed according to the usual recommendations: they will be given a diet and exercise plan in writing, which is the one commonly used in the Dietetics Unit, established by the Dietetics Unit according to patient age and level of activity, without any other assessment or additional visits by the Dietetics Unit. Visits to the Sleep Disorders Unit will be scheduled to coincide with the assessments at 3 and 12 months, the same as for the intervention group.

Criteria for withdrawal from the study:

* occurrence of osteoarticular pain that prevents a patient from continuing to exercise
* a patient's continued refusal to follow the recommended guidelines

RECRUITMENT PERIOD: Potential candidates will be selected from among patients who are being followed by their doctor or nurse for CPAP treatment. All potential candidates will be invited to participate in the study in consecutive order until the required number of patients has been reached.

MONITORING PERIOD: All patients will complete the one year of monitoring. If any adverse effects occur during the monitoring period, they will be recorded and discontinuation of the protocol will be assessed. Diet-related adverse effects are not expected as the patients will be followed very closely by the nutritionist. In the event any exercise-related osteoarticular pain should occur, the Rehabilitation Services will assess the patients and determine whether the exercise should be modified or discontinued.

ETHICAL ISSUES: The study will be conducted in accordance with the principles of the Declaration of Helsinki, as well as of the Data Protection Act (Law 15/1999). All patients will be asked to provide informed consent, in accordance with the rules of the Ethics Committee at our institution.

Since all of the patients will be receiving CPAP treatment, there should be no ethical concerns about evaluating the effectiveness of an alternative treatment that in principle is less effective than CPAP, in patients with severe OSAS.

STATISTICAL ANALYSIS:

In order to evaluate the effectiveness of a change in lifestyle (diet and exercise) in obese patients with OSAS, the investigators will first perform a descriptive analysis of the demographic variables and baseline characteristics according to the number of cases and percentages for the qualitative variables and the investigators will use measures of central tendency (mean, median) and dispersion (standard deviation and interquartile range) for the quantitative variables.

In order to answer the primary and secondary objectives of this study, the investigators will run an inferential analysis comparing data at baseline, at 3 months and at one year in the two treatment groups. Tests for independent samples will be used in every case (between the control and experimental groups). Either the chi-square test or Fisher's exact test will be used, as appropriate, to compare categorical variables and Student's T-test will be used to compare continuous variables; if the variable under study does not meet the conditions for the applicability of parametric tests, a non-parametric alternative, the Mann Whitney U test, will be used.

An estimate of treatment effect in answer to the primary and secondary endpoints will be obtained from the confidence interval (95% CI) of the difference between means and percentages, as appropriate.

Efficacy assessment will be based on an analysis of the per protocol populations (PP) and intention-to-treat (ITT), with ITT the population being the main analysis. For the population analysis using ITT, the missing data will be filled in and sensitivity analysis will be conducted if more than one method of imputation is used. The PP population will be determined in accordance with compliance with visits as well as with the diet and exercise.

A safety assessment will be made by identifying the adverse effects that are considered to be most significant due to their frequency or severity.

In all cases the significance level used will be 5% (α=0.05) with a bilateral approach.

The statistical software that will be used for the analysis will be International Business Machines Corporation (IBM) Statistical Package for the Social Sciences (SPSS) Statistics 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with severe obstructive sleep apnea syndrome (AHI > 30) and are already receiving CPAP treatment (since at least 6 months), who have class I and class II obesity (body mass index (BMI) >= 30 kg /m2 y <= 40 kg/m2).

Exclusion Criteria:

* diseases that limit exercising or diet,
* cognitive impairment that prevents understanding the program,
* psychiatric disorders,
* severe diseases, major cardiovascular disease,
* clinical instability within the previous month,
* prior bariatric surgery,
* refusal to participate in the study,
* participation in another clinical trial.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Improvement in the apnea-hypopnea index/hour: Sleep study: Standard polysomnography | Baseline, at 3 months and 12 months.
  Assess whether a lifestyle change program can be effective in the medium and long term for the treatment of OSAS in obese patients with OSAS who are already receiving CPAP treatment.

SECONDARY OUTCOMES:
waist circumference (above the upper iliac crest): centimetre | Baseline, at 3 months and 12 months.
neck circumfarence: centimetre | Baseline, at 3 months and 12 months.
waist to hip ratio | Baseline, at 3 months and 12 months.
Measurement of visceral fat (square centimetre) by an abdominal computerized tomography (CT) scan | Baseline, at 12 months.
Carotid intima-media (C-IMT) thickness (millimeter (mm)) by ultrasound of the supra-aortic vessels, using B-mode ultrasound | Baseline, at 3 months and 12 months.
  As a marker of subclinical cardiovascular disease
Body fat composition by bioimpedance analysis (BIA 101, Akern Bioresearch, Florence, Italy). | Baseline, at 3 months and 12 months.
Measurement of health-related quality of life | Baseline, at 3 months and 12 months.
  Questionnaire regarding quality of life and sleep: Functional Outcomes of Sleep Questionnaire (FOSQ), Spanish language version (Ferrer et al Med Clin (Barc 1999; 113: 250-5).
Measurement of health-related quality of life | Baseline, at 3 months and 12 months.
  Self-administered questionnaire regarding quality of life and sleep-related breathing disorders: Quebec Sleep Questionnaries (QSQ), Spanish language version (Lacasse et al Thorax 2004; 59: 494-9).
Measurement of health-related quality of life | Baseline, at 3 months and 12 months.
  Euro quality of life (EuroQol) and the Analog pain scale for the assessment of well-being with regard to the disease under study. (Masa et al AJRCCM 2004 and Sleep and Breathing 2011).
Age (years) | Baseline, at 3 months and 12 months.
Self-perceived sleepiness | Baseline, at 3 months and 12 months.
  It will be analyzed using the Epworth Sleepiness Scale (MW Johns, Sleep 1991, 14;540).
Cardiovascular risk factors and comorbidity. | Baseline, at 3 months and 12 months.
  Using general medical history questionnaire
OSAS-related symptoms | Baseline, at 3 months and 12 months.
Testing for ketones (milligram/deciliter) using test strips | Baseline, at 3 months and 12 months.
Record of physical activity: hours of exercise will be noted daily in a journal | Baseline, at 3 months and 12 months.
Exercise capacity: 6 minute walk test (6MWT) | Baseline, at 3 months and 12 months.
Pain: VAS Analog Scale for Pain | Baseline, at 3 months and 12 months.
Blood pressure | Baseline, at 3 months and 12 months.
CPAP compliance (mean hours of usage per night as recorded by the hour meters). | Baseline, at 3 months and 12 months.
CPAP related side effects | Baseline, at 3 months and 12 months.
Hours of sleep | Baseline, at 3 months and 12 months.
Fibrinogen (gram/liter) | Baseline, at 3 months and 12 months.
Glucose (millimole/liter) | Baseline, at 3 months and 12 months.
Markers of endothelial dysfunction: Asymetric Dimethylarginine (ADMA), intercellular adhesion molecule (ICAM-1), vascular endothelial cell adhesion molecule (VCAM-1), vascular endothelial growth factor (VEGF), endothelin | Baseline, at 3 months and 12 months.
Platelet activation and markers of the fibrinolytic system: p-selectin, Soluble CD40 ligand (sCD40), Plasminogen activator inhibitor (PAI-1) | Baseline, at 3 months and 12 months.
Markers of hemodynamic dysfunction: N-terminal pro brain natriuretic peptide (NT-proBNP) | Baseline, at 3 months and 12 months.
Markers of oxidative stress: isoprostanes | Baseline, at 3 months and 12 months.
Markers of inflammation: interleukin (IL) 6, IL-8, tumor necrosis factor (TNF) alpha and TNF soluble receptors 1 and 2, adiponectin | Baseline, at 3 months and 12 months.
Gender: male, female | Baseline
Weight (kilograme) | Baseline, at 3 months, and 12 months.
Height (meter) | Baseline, at 3 months, and 12 months.
Body mass index (BMI): dividing weight in kilograms by height in meters squared | Baseline, at 3 months, and 12 months.
Start of Obesity: period of obesity | Baseline
Adherence to diet monitoring by diet questionnaries | Baseline, at 3 months and 12 months
D-dimer (microgram/liter) | Baseline, at 3 months and 12 months
Prothrombin time (PT) | Baseline, at 3 months and 12 months
Activated partial thrombopastin time (APTT) | Baseline, at 3 months and 12 months
Triglycerides (millimole/liter) | Baseline, at 3 months and 12 months
Total cholesterol (millimole/liter) | Baseline, at 3 months and 12 months
Low density lipoprotein (LDL) cholesterol (millimole/liter) | Baseline, at 3 months and 12 months
High density lipoprotein (LDL) cholesterol (millimole/liter) | Baseline, at 3 months and 12 months
Uric acid (micromole/liter) | Baseline, at 3 months and 12 months
Creatinine (micromole/liter) | Baseline, at 3 months and 12 months
C-reactive protein (milligram/liter) | Baseline, at 3 months and 12 months
Aspartate aminotransferase (microgram/liter) | Baseline, at 3 months and 12 months
Alanine aminotransferase (microgram/liter) | Baseline, at 3 months and 12 months
Thyroid-Stimulating Hormone (TSH) | Baseline, at 3 months and 12 months
Glycosylated hemoglobin | Baseline, at 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Monasterio Ponsa, Doctor, Principal Investigator — Hospital Universitari Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Lopez-Padros C, Salord N, Alves C, Vilarrasa N, Gasa M, Planas R, Montsserrat M, Virgili MN, Rodriguez C, Perez-Ramos S, Lopez-Cadena E, Ramos MI, Dorca J, Monasterio C. Effectiveness of an intensive weight-loss program for severe OSA in patients undergoing CPAP treatment: a randomized controlled trial. J Clin Sleep Med. 2020 Apr 15;16(4):503-514. doi: 10.5664/jcsm.8252. PMID 32003737